CLINICAL TRIAL: NCT03742531
Title: Does Induction Dosage in Latent Phase Affect Active Phase of Labor?A Randomized Study
Brief Title: Does Induction Dosage in Latent Phase Affect Active Phase of Labor?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, principal investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50
Record Dates: First submitted 2018-03-25; First posted 2018-11-15 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Oxytocin; Induction of Labor
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- low dose group (Active Comparator): oxytocin therapy starting with 2mU/min increased by 2 mU/min every 15 minutes. oxytocin will be stopped at the beginning of the active phase of labor.
  Interventions: Drug: oxytocin
- high dose group (Active Comparator): oxytocin therapy starting with 4mU/min increased by 4 mU/min every 15 minutes. oxytocin will be stopped at the beginning of the active phase of labor.
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — one group will be treated with low dose oxytocin and the other group will be treated with high dose oxytocin for augmentation of labor induction.
  Other Names: synpitan

SUMMARY:
This study evaluates the need of oxytocin therapy in active phase of labor. there will be two groups treating with oxytocin in latent phase.One group will be treated with low dose oxytocin therapy and the other group will be treated with high dose oxytocin therapy. oxytocin treatment will be ceased at the beginning of the active phase of labor. the need of oxytocin treatment in active phase of labor will be compared between two groups.

DETAILED DESCRIPTION:
Oxytocin treatment in active phase of labour is used with respect to clinicians preference and best approach has not been described. We want to investigate the effect of oxytocin treatment by using different regims in latent phase of labor when oxytocin treatment is ceased in active phase of labour. In our trial we discontinued oxytocin in active phase of labour and investigate which group needs oxytocin therapy due to inadequate uterine contractions and arrest of labor.

ELIGIBILITY:
Inclusion Criteria:

* Live fetus in cephalic presentation, sonographically estimated fetal weight less than 4200 g, undergoing induction of labor at 37-42 weeks of gestation, having indications of labor, no previous uterine surgery

Exclusion Criteria:

* malpresentation, placenta previa, previous uterine surgery, multiple gestation, active genital herpes, non-reassuring fetal heart rate pattern

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — term pregnant women
Enrollment: 300 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
need for oxytocin retreatment | an average of one year
  need for oxytocin retreatment due to inadequate uterine contractions and labor arrest

SECONDARY OUTCOMES:
length of active phase | an average of one year
  duration of acive phase of labor
ratio of caesarean section | an average of one year
  caesaraen section rate in total delivery
total oxytocin dose | an average of one year
  total amount of oxytocin treatment in latent and active phase of labor
APGAR scores | an average of one year
  neonatal 1 minute and 5-minute-APGAR scores

CONTACTS AND LOCATIONS:
Overall Officials: ahmet eser, Principal Investigator — Zeynep Kamil Education and Research Hospital
Locations (1):
- Zeynep Kamil Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided